CLINICAL TRIAL: NCT06081023
Title: Development and Feasibility of Psycho-Educational Weight Reduction Program for Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: 2020(fall).MPhil(Psy)-009
Record Dates: First submitted 2023-04-12; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Emotional Eating; Obesity
Keywords: Psycho-educational weight reduction program
MeSH Terms: conditions — Emotional Eating; Obesity

STUDY DESIGN:
Intervention Model Description: Two groups i-e control and experimental. The experimental group was provided with treatment while the control group was only provided with behavioral relaxing techniques.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (No Intervention): This arm was provided with only a relaxing behavioral technique
- Psycho-educational weight reduction program (Experimental): This arm was provided with treatment of reducing emotional eating and obesity level
  Interventions: Behavioral: Psycho-educational weight reduction program

INTERVENTIONS:
Behavioral: Psycho-educational weight reduction program — This program provides behavioral technique in order to minimize level of emotional eating and level of obesity
  Arms: Psycho-educational weight reduction program

SUMMARY:
The main aim of the study was to assess the efficacy of psycho-educational weight reduction program for reducing emotional eating and obesity

DETAILED DESCRIPTION:
All participants who provide written informed consent will go through a screening process to evaluate their eligibility for study entrance after being briefed about the study and any potential risks. Individuals who met the eligibility requirements will then be randomly assigned to the control group and the experimental group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be enrolled at a university.
* Based on World Health Organizations age range young adults were selected for the current study i-e 19 years to 35 years (WHO; 2019).

Exclusion Criteria:

* The young adults who diagnosed with any chronic health concern, either psychological or physical must not be included in the current study.
* The individuals who joined any kind of weight loss program or gym were also not included in the study.
* Individuals older than 35 were not included in the current study either.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Emotional Eating on Emotional Eating Scale (EES-25) after 12 weeks | Baseline and Week 12
  The EES-25 is a validated self-report scale assessing the level of emotional eating. Possible scores range from 25 (No desire to eat) to 125 (an overwhelming urge to eat) Change=week 12 score-baseline score

CONTACTS AND LOCATIONS:
Locations (1):
- Nimra Anjum, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All the obtained information will be shared maintaining confidentiality and anonymity of obtained data
Supporting Information: Study Protocol, SAP, ICF, CSR